CLINICAL TRIAL: NCT05157815
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Investigate the Effect of 16 Weeks of Twice Daily Supplementation With Soluble Corn Fibre on Long Term Glucose Control in Prediabetic Subjects
Brief Title: Study to Investigate the Effect of Dietary Fibre Supplementation on Long-term Glucose Control in Prediabetic Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tate & Lyle (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry); University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AFCRO-129
Record Dates: First submitted 2021-11-16; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Dietary Habits
Keywords: glycemia; fiber; prediabetes
MeSH Terms: conditions — Feeding Behavior; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind: The relationship between the randomisation number and the group assignment will be unknown to the clinical research team, the sponsor, trial site staff, and the participants, i.e. the trial will be double-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soluble Corn Fibre (Experimental): 12g compound per Sachet (providing 10g fibre) consumed twice per day
  Interventions: Dietary Supplement: Soluble Fibre
- Maltodextrin (Placebo Comparator): Calorie matched control of 2 g compound per sachet (0 g fibre), composed of: Maltodextrin, consumed twice per day
  Interventions: Dietary Supplement: Calorie Matched Control

INTERVENTIONS:
Dietary Supplement: Soluble Fibre — 10g soluble corn fibre to be consumed twice per day
  Arms: Soluble Corn Fibre
Dietary Supplement: Calorie Matched Control — 2g maltodextrin consumed twice per day
  Arms: Maltodextrin

SUMMARY:
The purpose of the study is to explore the potential metabolic health benefits of a dietary fibre intervention by using Soluble Fibre in a human intervention study in Healthy Obese Pre-diabetic participants over a period of 16 weeks with a focus on long term glucose control.

The hypothesis is that twice daily supplementation with Soluble Fibre over a period of 16 weeks will significantly improve long term glucose control in pre-diabetic participants.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Males & females aged 18 to 70 years (inclusive).
3. Has a BMI between ≥30 and ≤40 kg/m2.
4. HbA1c between ≥38.8 and ≤47 mmol/mol (5.7-6.4 %)
5. Has a stable body weight (≤5 % change) over the past 3-months.
6. Is in general good health, as determined by the investigator.
7. Willing to consume the investigational product daily for the duration of the trial.
8. Willing to wear a continuous glucose monitoring sensor for two 14-day periods.
9. Be willing to maintain stable dietary habits and physical activity levels throughout the trial period.

Exclusion Criteria:

* 1. Are aged less than 18 or greater than 70 years. 2. Participants who are pregnant, breastfeeding, or wish to become pregnant during the trial.

  3. Participants currently of childbearing potential, but not using an effective method of contraception, as outlined below:
  1. Complete abstinence from intercourse two weeks prior to administration of the investigational product, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the investigational product in cases where participant discontinues the trial prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit).
  2. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that participant.
  3. Sexual partner(s) is/are exclusively female.
  4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm) or contraceptive pill. The participant must be using this method for at least 1 week following the end of the trial.
  5. Use of any non-hormonal intrauterine device (IUD) or contraceptive implant with published data showing that the highest expected failure rate is less than 1 % per year. The participant must have the device inserted at least 2 weeks prior to the first Screening Visit, throughout the trial, and 2 weeks following the end of the trial.

     4. Are hypersensitive to any of the components of the investigational product or common food allergens.

     5. Has taken antibiotics within the previous 12-weeks prior to randomisation 6. Participant regularly takes probiotics, prebiotics, or fibre supplements (daily use in the 4 weeks prior to screening and up to baseline) 7. Has an intake of more than 19 g of fibre per day. 8. Has taken anti-obesity medication/supplement within the previous 12-weeks prior to randomisation.

     9. Participant is actively or has recently (3 months prior to randomisation) participated in a weight loss program or weight change of 5 % during the past 3 months.

     10. Participant has Type 1 or Type 2 Diabetes Mellitus. 11. Has a history of bariatric surgery. 12. Participant who is severely immuno-compromised (HIV positive, transplant patient, on antirejection medications, or has undergone chemotherapy or radiotherapy within the last year).

     13. Participant has significant comorbidities or an uncontrolled disease, as determined by the PI/Sub-Investigator on the basis of medical history and routine laboratory test results that may adversely affect the participant's ability to complete the trial or it's assessments or which may pose significant risk to the participant.

     14. Participant has a history of co-existing gastrointestinal, and/or gynaecological, and/or urologic pathology (e.g., colon cancer, colitis, Crohn's Disease, Celiac, Endometriosis, prostate cancer) or lactose intolerance.

     15. Has a gastrointestinal or chronic infective disease (i.e., diarrhoea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, HIV, cancer, etc.), or with a history of such diseases.

     16. Has a history of drug and/or alcohol abuse at the time of enrolment.

  <!-- -->

  1. Consumes greater than nationally recommended units of alcohol per week (>11 units for women & >17 units for men).
  2. Is currently in treatment (or has been in the last 6 months) for alcohol/substance abuse
  3. Has been diagnosed with alcohol/substance abuse disorder. 17. Has used oral/injectable steroids within the previous 30 days prior to Screening (or between Screening/Baseline Visit).

     18. Taking a medication that the investigator believes would interfere with the objectives of the trial or pose a safety risk or confound the interpretation of the trial results. Prohibited medications include:

  <!-- -->

  1. Metformin
  2. Anti-psychotic drugs 19. If taking anti-hypertensive drugs, anti-depressive drugs, statins, or any other medication that the investigator determines could impact the results of the study, the participant must have been taking the product for at least 3 months prior to screening. (Changes to the dose during the trial will be assessed by the investigator for impact on trial results).

     20. Individual who work a shift work pattern that requires them to work >1 nightshift per week.

     21. Individuals living in the same residence as a previously or currently enrolled participants on the trial.

     22. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.

     23. Participant is currently, or planning, to participate in another interventional study during the study period.

     24. Participants may not be receiving treatment involving experimental drugs. If the participant has been in a recent experimental trial, these must have been completed not less than 30 days prior to this trial.

     25. Individuals who have a history of non-compliance or, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in plasma HbA1c concentration | 16 weeks
  Change from baseline to week 16 in the treatment group compared to placebo on plasma HbA1c (mmol/mol) concentration

SECONDARY OUTCOMES:
Change in post-prandial Blood Glucose (mmol/L) measured by incremental Area Under the Curve (iAUC) derived from an Oral Glucose Tolerance Test (OGTT) | 16 weeks
Change in post-prandial Blood Glucose maximal concentration, derived from an Oral Glucose Tolerance Test (OGTT) | 16 weeks
Change in post-prandial Blood Glucose time to peak, derived from an Oral Glucose Tolerance Test (OGTT) | 16 weeks
Change in post-prandial insulin (mIU/L) as measured by incremental Area Under the Curve (iAUC) derived from an Oral Glucose Tolerance Test (OGTT) | 16 weeks
Change in post-prandial insulin maximal concentration (Cmax) derived from an Oral Glucose Tolerance Test (OGTT) | 16 weeks
Change in post-prandial Blood Insulin time to peak (Tmax), derived from an Oral Glucose Tolerance Test (OGTT) | 16 weeks
Change in insulin resistance (mIU/L) | 16 weeks
Change in lipids (mmol/L): Triglycerides (TG), Total Cholesterol (TC), High-Density Lipoprotein Cholesterol (HDL), Low-Density Lipoprotein Cholesterol (LDL) | 16 weeks
Change in waist-to-hip ratio | 16 weeks
Change in BMI (kg/m2) | 16 weeks
Continuous blood glucose monitoring (during run-in & 2-weeks before End of Study) as measured by Freestyle Libre Glucose Monitoring System, a continuous glucose monitoring (CGM) device. | 16 weeks
Change in Fasting Blood Glucose (FBG) (mmol/L) | 16 weeks
Change in Fasting Insulin (mIU/L). | 16 weeks

OTHER OUTCOMES:
Change in gut hormones (GLP-1 and PYY) measured by iAUC (T-15 to T120 minutes) | 16 weeks
Change in self-reported hunger and satiety measured by iAUC (T-15 to T120 minutes) | 16 weeks
Change in the composite score of gastrointestinal symptoms, (bloating score + abdominal cramping score + stomach noises score + flatulence score) | 16 weeks
Change in stool consistency (Bristol Stool Scale) and frequency | 16 weeks
Change in Faecal Short Chain Fatty Acids (fSCFA) microbiota | 16 weeks
Change in TNF alpha | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No